CLINICAL TRIAL: NCT06435780
Title: Evaluation of a Novel Technique Versus Conventional Subepithelial Connective Tissue Graft in Treatment of Ridge Contour Defects. A Randomized Controlled Clinical Trial
Brief Title: Novel Technique Versus Conventional Subepithelial Connective Tissue Graft in Treatment of Ridge Contour Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Clinical Director of International Implantology Program (IIP), Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWA #00022887
Record Dates: First submitted 2024-02-04; First posted 2024-05-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Defect in Alveolar Ridge
Keywords: ridge contour defect; soft tissue graft; Rolling Technique; Connective tissue graft; Subepithelial palatal graft; Seibert Class I

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Augmentation of soft tissue by a novel Denuded interpositional pedicled rolled flap technique (DIPRF)
  Interventions: Procedure: DIPRF
- Control group (Active Comparator): Will be augmented by the conventional subepithelial connective tissue graft technique.
  Interventions: Procedure: DIPRF

INTERVENTIONS:
Procedure: DIPRF — Denuded interpositional pedicled rolled flap technique

SUMMARY:
The aim of the study is to clinically and radiographically evaluate and compare two techniques to augment soft tissues: the conventional subepithelial connective tissue graft technique and a novel denuded interpositional pedicled rolled flap technique (DIPRF) These techniques will be used to augment edentulous ridges that are recommended for rehabilitation by an implant or a fixed restoration.

DETAILED DESCRIPTION:
Fifty patients with soft tissue ridge contour defects in the maxillary premolar region and recommended for rehabilitation by an implant or a fixed restoration will be enrolled. Patients will be allocated randomly into two groups; group 1 (test group) will have augmentation for their soft tissue by a novel Denuded interpositional pedicled rolled flap technique (DIPRF); group 2 (control group) will be augmented by the conventional subepithelial connective tissue graft technique. Clinical volumetric change evaluation and ridge thickness analysis using digitally calibrated casts and CBCT analysis with a fusion software will be performed for every site as well as periodontal evaluation and patient centered outcomes, including pain and satisfaction after the procedure will be recorded for both techniques. For each site, an impression will be used to pour a cast that will be digitally scanned and vertical and horizontal ridge contours dimensions(tissue volumetric changes) will be recorded. These measurements will be obtained before the surgical procedure, 2 weeks, and 3 and 6 months post-surgical. CBCT analysis will be performed pre-operatively to confirm the diagnosis and eligibility of the case as having only soft tissue defect without bone defects, and 6 months postoperatively to analyze the amount of soft tissue gain in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adults above the age of 18 to 50 years.
2. Males and females as confirmed by asking the female patients about whether they are pregnant or not
3. Patient's with Seibert classification class I requiring future rehabilitation of one or more premolar region and sound adjacent teeth.
4. Soft tissue thickness on the palatal tissues more than 6mm at the site of harvesting the graft.
5. Presence of Mandibular posterior teeth opposing the tooth to be replaced for occlusion.
6. Clinically healthy soft tissues with no signs of clinical pathology of the soft tissue.
7. Good oral hygiene.
8. Patient accepts to sign an informed consent.
9. ASA I or ASA II Patient.

Exclusion Criteria:

1. Patients with ridge defects due to bone defect
2. Smoker patients who smoke more than 10 cigarettes per day
3. Pregnant females

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ridge contour thickness gain | 6 months
  Ridge contour will be assessed using CBCT analysis using fusion software. The differences between measurement times will indicate the amount of bone gain

CONTACTS AND LOCATIONS:
Overall Officials: Hebattallah A Mattar, Principal Investigator — Misr International University
Locations (1):
- Misr International University, Cairo, Egypt

REFERENCES:
- [Background] Scharf DR, Tarnow DP. Modified roll technique for localized alveolar ridge augmentation. Int J Periodontics Restorative Dent. 1992;12(5):415-25. PMID 1343013
- [Background] Su H, Gonzalez-Martin O, Weisgold A, Lee E. Considerations of implant abutment and crown contour: critical contour and subcritical contour. Int J Periodontics Restorative Dent. 2010 Aug;30(4):335-43. PMID 20664835
- [Background] Seibert JS. Reconstruction of deformed, partially edentulous ridges, using full thickness onlay grafts. Part I. Technique and wound healing. Compend Contin Educ Dent (Lawrenceville). 1983 Sep-Oct;4(5):437-53. No abstract available. PMID 6578906
- [Background] Meltzer JA. Edentulous area tissue graft correction of an esthetic defect. A case report. J Periodontol. 1979 Jun;50(6):320-2. doi: 10.1902/jop.1979.50.6.320. PMID 287786
- [Background] Langer B, Calagna L. The subepithelial connective tissue graft. J Prosthet Dent. 1980 Oct;44(4):363-7. doi: 10.1016/0022-3913(80)90090-6. PMID 6931898
- [Background] Kaldahl WB, Tussing GJ, Wentz FM, Walker JA. Achieving an esthetic appearance with a fixed prosthesis by submucosal grafts. J Am Dent Assoc. 1982 Apr;104(4):449-52. doi: 10.14219/jada.archive.1982.0209. PMID 6950973
- [Background] Garber DA, Rosenberg ES. The edentulous ridge in fixed prosthodontics. Compend Contin Educ Dent (Lawrenceville). 1981 Jul-Aug;2(4):212-23. No abstract available. PMID 6950860
- [Background] Abrams L. Augmentation of the deformed residual edentulous ridge for fixed prosthesis. Compend Contin Educ Gen Dent. 1980 May-Jun;1(3):205-13. No abstract available. PMID 6950834
- [Background] Soehren SE, Allen AL, Cutright DE, Seibert JS. Clinical and histologic studies of donor tissues utilized for free grafts of masticatory mucosa. J Periodontol. 1973 Dec;44(12):727-41. doi: 10.1902/jop.1973.44.12.727. No abstract available. PMID 4586681
- [Background] Akcali A, Schneider D, Unlu F, Bicakci N, Kose T, Hammerle CH. Soft tissue augmentation of ridge defects in the maxillary anterior area using two different methods: a randomized controlled clinical trial. Clin Oral Implants Res. 2015 Jun;26(6):688-95. doi: 10.1111/clr.12368. Epub 2014 Apr 10. PMID 24720375
- [Background] Mormann W, Schaer F, Firestone AR. The relationship between success of free gingival grafts and transplant thickness. Revascularization and shrinkage--a one year clinical study. J Periodontol. 1981 Feb;52(2):74-80. doi: 10.1902/jop.1981.52.2.74. PMID 6164778
- [Background] Studer SP, Lehner C, Bucher A, Scharer P. Soft tissue correction of a single-tooth pontic space: a comparative quantitative volume assessment. J Prosthet Dent. 2000 Apr;83(4):402-11. doi: 10.1016/s0022-3913(00)70034-5. PMID 10756289
- [Background] Thoma DS, Benic GI, Zwahlen M, Hammerle CH, Jung RE. A systematic review assessing soft tissue augmentation techniques. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:146-65. doi: 10.1111/j.1600-0501.2009.01784.x. PMID 19663961
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Gurlek O, Sonmez S, Guneri P, Nizam N. A novel soft tissue thickness measuring method using cone beam computed tomography. J Esthet Restor Dent. 2018 Nov;30(6):516-522. doi: 10.1111/jerd.12428. Epub 2018 Nov 15. PMID 30444040
- [Background] Das G, Ahmed AR, Suleman G, Lal A, Rana MH, Ahmed N, Arora S. A Comparative Evaluation of Dentogingival Tissue Using Transgingival Probing and Cone-Beam Computed Tomography. Medicina (Kaunas). 2022 Sep 19;58(9):1312. doi: 10.3390/medicina58091312. PMID 36143989
- [Background] Smeets EC, de Jong KJ, Abraham-Inpijn L. Detecting the medically compromised patient in dentistry by means of the medical risk-related history. A survey of 29,424 dental patients in The Netherlands. Prev Med. 1998 Jul-Aug;27(4):530-5. doi: 10.1006/pmed.1998.0285. PMID 9672946
- [Background] Ammar AH, Ahmed E, ElBarbary A, Ghalwash D, Ezz Elarab A. Clinical Comparison of the Volumetric Changes in Single Pontic Site Development through Connective Tissue Grafting Using Modified Pouch Technique versus Pouch Technique in the Maxillary Esthetic Zone: A Randomized Controlled Clinical Trial. Int J Dent. 2022 Aug 25;2022:1677471. doi: 10.1155/2022/1677471. eCollection 2022. PMID 36059913